CLINICAL TRIAL: NCT07220044
Title: Effects of Streak-Based Versus Tally-Based Feedback on Daily Lesson Completion During a 30-Day Digital Health Challenge
Acronym: Streaks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DBSR-11288; P30AG034546-16 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Preventive Health Care
Keywords: Behavioral Science; Field Experiment; Streaks
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streaks (Experimental): In the streak group, participants would see how many consecutive days they have completed daily lessons and will be encouraged to extend their streak
  Interventions: Behavioral: Interventions for increasing engagement with a target behavior
- Tally (Experimental): In the tally group, participants will see how many cumulative days they have completed daily lessons and will be encouraged to extend their tally.
  Interventions: Behavioral: Interventions for increasing engagement with a target behavior

INTERVENTIONS:
Behavioral: Interventions for increasing engagement with a target behavior — The study will test two interventions for increasing engagement with a target behavior, delivered via a digital web application that participants can access using their phones or computers. For example, in the streak group, participants would see how many consecutive days they have completed daily lessons and will be encouraged to extend their streak. In the tally group, participants will see how many cumulative days they have completed daily lessons and will be encouraged to extend their tally. The investigators are interested in whether people complete more daily lessons when a 30-day health challenge app provides daily feedback on their consecutive lessons (each comprising two multiple-choice questions) completed (i.e., "streaks") vs. when it provides feedback on their cumulative lessons completed (i.e., "tallies").

SUMMARY:
The study will test two interventions for increasing engagement with a target behavior, delivered via a digital web application that participants can access using their phones or computers. For example, in the streak group, users would see how many consecutive days they have completed daily lessons and will be encouraged to extend their streak. In the tally group, participants will see how many cumulative days they have completed daily lessons and will be encouraged to extend their tally.

DETAILED DESCRIPTION:
The objective of this study is to determine whether tracking people's streak of behavior increases their engagement in that behavior. To test this, the investigators are designing a web application that participants can access daily using their phones or computers. Our previous work suggests that streaks may be useful in motivating people to be more productive. In this study, the investigators change how the investigators operationalize streaks and test streaks in a field context. Because most previous streak research is on how others perceive someone who has a streak, this work is novel because it examines how encouraging someone to achieve and keep a streak affects behavior in a field context. The study will test two interventions for increasing engagement with a target behavior, delivered via a digital web application that participants can access using their phones or computers. For example, in the streak group, users would see how many consecutive days they have completed daily lessons and will be encouraged to extend their streak. In the tally group, participants will see how many cumulative days they have completed daily lessons and will be encouraged to extend their tally. The investigators are interested in whether people complete more daily lessons when a 30-day health challenge app provides daily feedback on their consecutive lessons (each comprising two multiple-choice questions) completed (i.e., "streaks") vs. when it provides feedback on their cumulative lessons completed (i.e., "tallies").

ELIGIBILITY:
Inclusion Criteria:

* Our target population is 18 and older adults in the United States who have a valid U.S. phone number and who are willing to make an account on our web application for use during the duration of the study.

Exclusion Criteria:

* Children under 18 years of age and adults without a valid U.S. phone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7004 (Actual)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Total number of lessons completed | 30 days
  The key dependent variable is a person's total number of lessons completed during the 30-day Health Daily program. Participants can only complete a given day's lesson on that day; a lesson is only considered complete if both questions that comprise the lesson are answered.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
* Unique ID
  * Condition assignment
  * Response for the first quiz question for each day
  * Response for the second quiz question for each day
  * Date
  * Female indicator (taken from generize.io)
  * Correct response for the first quiz question
  * Correct response for the second quiz question
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Individual participant data and all supporting materials will become available upon publication of the primary study manuscript and will remain accessible indefinitely thereafter.
Access Criteria: Individual participant data and all supporting materials will be made openly available through the Open Science Framework (OSF) to any interested party without access restrictions.
URL: https://osf.io/e3w7t/overview?view_only=6846fba28326480ca8742041dac10247